CLINICAL TRIAL: NCT02969408
Title: A 12-Week, Open-Label Study to Evaluate the Relationship Between Use of Albuterol eMDPI, an Inhaled Short-Acting Beta Agonist "Rescue" Agent With an eModule, and Exacerbations in Patients (18 Years of Age or Older) With Asthma
Brief Title: A Study to Evaluate the Relationship Between Use of Albuterol Multidose Dry Powder Inhaler With an eModule (eMDPI) and Exacerbations in Participants With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABS-AS-30064
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABS eMDPI (Experimental): Participants will receive 90 mcg of ABS via an eMDPI (sitting on the upper part of the device for the purposes of detecting and storing usage information), 1 to 2 inhalations every 4 hours, as needed for 12 weeks.
  Interventions: Drug: Albuterol Sulfate

INTERVENTIONS:
Drug: Albuterol Sulfate — Albuterol sulfate will be administered as per the dose and schedule specified in the arm.

SUMMARY:
This is a Phase 3B, 12-week, multicenter, open-label study to evaluate the relationship between albuterol sulfate (ABS) eMDPI and clinical asthma exacerbation (CAE) in adult participants at least 18 years of age with exacerbation-prone asthma. The ABS eMDPI dose will be 90 micrograms (mcg), 1 to 2 inhalations every 4 hours as needed, but participant dosing will not be limited to this dosing regimen. The purpose of this study is to evaluate the relationship between albuterol dosing and CAE.

ELIGIBILITY:
Inclusion Criteria:

* The participant has had at least 1 episode of a severe CAE over the past 12 months before screening. If on a biologic (for example, omalizumab, mepolizumab, or reslizumab) and/or post-bronchial thermoplasty, exacerbation has occurred after these interventions.
* The participant is using a moderate-dose inhaled corticosteroid (ICS) equivalent to at least 440 mcg daily of fluticasone propionate.
* The participant's baseline asthma therapy regimen, including oral corticosteroids, leukotriene antagonists, 5-lipoxygenase inhibitors, long-acting beta agonist (LABA), long-acting muscarinic agent, or cromolyn, biologicals, theophylline, or mepolizumab, is allowed.
* The participant must be willing and able to comply with study requirements as specified in the protocol, including the use of a wearable accelerometer for the subset of participants who consent to use of the device.
* The participant is willing to discontinue all other rescue or maintenance short-acting beta 2 agonist (SABA) or antimuscarinic agents and replace them with the study-provided ABS eMDPI for the duration of the trial.
* Women of childbearing potential (not surgically sterile or at least 2 years postmenopausal) must have exclusively same-sex partners or use a highly effective method of birth control and must agree to continue the use of this method for the duration of the study and for 30 days after discontinuation of the investigational medicinal product (IMP).

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has any clinically significant medical condition (treated or untreated) that, in the opinion of the investigator, would interfere with participation in the study.
* The participant has any other confounding underlying lung disorder other than asthma.
* The participant has used an investigational drug within 5 half-lives of it being discontinued or 1 month of baseline visit, whichever is longer.
* The participant is a pregnant or lactating woman, or plans to become pregnant during the study. Note: Any woman becoming pregnant during the study will be withdrawn from the study.
* The participant is known to be allergic to albuterol or any of the excipients in the IMP or rescue medication formulation (that is, lactose). Dietary lactose intolerance does not exclude the participant from inclusion in the study or as per the investigator's medical discretion.
* The participant has a history or presence of "silent" infections, including positive testing for human immunodeficiency virus types 1 and 2, hepatitis B, hepatitis C, and tuberculosis.

  * Additional criteria apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (44):
- United States (44):
  - Teva Investigational Site 13964, Litchfield Park, Arizona
  - Teva Investigational Site 13959, Bakersfield, California
  - Teva Investigational Site 13954, Los Angeles, California
  - Teva Investigational Site 13923, Orange, California
  - Teva Investigational Site 13961, Riverside, California
  - Teva Investigational Site 13933, Centennial, Colorado
  - Teva Investigational Site 13946, Clearwater, Florida
  - Teva Investigational Site 13921, Loxahatchee Groves, Florida
  - Teva Investigational Site 13942, Miami, Florida
  - Teva Investigational Site 13927, Miami, Florida
  - Teva Investigational Site 13948, Orlando, Florida
  - Teva Investigational Site 13934, Orlando, Florida
  - Teva Investigational Site 13931, Ormond Beach, Florida
  - Teva Investigational Site 13926, Sarasota, Florida
  - Teva Investigational Site 13963, Savannah, Georgia
  - Teva Investigational Site 13943, Michigan City, Indiana
  - Teva Investigational Site 13925, Overland Park, Kansas
  - Teva Investigational Site 13958, Fort Mitchell, Kentucky
  - Teva Investigational Site 13940, Owensboro, Kentucky
  - Teva Investigational Site 13937, Bangor, Maine
  - Teva Investigational Site 13965, St Louis, Missouri
  - Teva Investigational Site 13919, Missoula, Montana
  - Teva Investigational Site 13947, Bellevue, Nebraska
  - Teva Investigational Site 13960, Brick, New Jersey
  - Teva Investigational Site 13932, Piscataway, New Jersey
  - Teva Investigational Site 13922, Verona, New Jersey
  - Teva Investigational Site 13945, Rochester, New York
  - Teva Investigational Site 13936, High Point, North Carolina
  - Teva Investigational Site 13953, Cincinnati, Ohio
  - Teva Investigational Site 13928, Edmond, Oklahoma
  - Teva Investigational Site 13955, Oklahoma City, Oklahoma
  - Teva Investigational Site 13949, East Providence, Rhode Island
  - Teva Investigational Site 13929, Charleston, South Carolina
  - Teva Investigational Site 13941, Greenville, South Carolina
  - Teva Investigational Site 13951, Greenville, South Carolina
  - Teva Investigational Site 13938, Spartanburg, South Carolina
  - Teva Investigational Site 13924, Knoxville, Tennessee
  - Teva Investigational Site 13962, Boerne, Texas
  - Teva Investigational Site 13920, Dallas, Texas
  - Teva Investigational Site 13930, Houston, Texas
  - Teva Investigational Site 13939, San Antonio, Texas
  - Teva Investigational Site 13957, San Antonio, Texas
  - Teva Investigational Site 13952, South Burlington, Vermont
  - Teva Investigational Site 13956, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 449 participants with exacerbation-prone asthma were screened, of which 397 participants at 45 investigational centers in the US met entry criteria and were considered to be eligible for enrollment into the study.
Groups:
- ABS eMDPI: Participants received 90 micrograms (mcg) of albuterol sulfate (ABS) via a multidose dry powder inhaler (MDPI) with an eModule (eMDPI) (sitting on the upper part of the device for the purposes of detecting and storing usage information), 1 to 2 inhalations every 4 hours, as needed for 12 weeks. ABS eMDPI was a rescue/reliever agent that included an eModule on top of the approved PROAIR RESPICLICK® inhaler. Participants were allowed to continue use of other asthma and non-asthma medications as advised by their physician without changes unless deemed necessary by their physician.
Period: Overall Study
Arm/Group | ABS eMDPI
Started | 397
Used ABS eMDPI at Least Once | 370
Completed | 381
Not Completed | 16
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 1
Not completed — Other than specified | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all enrolled participants regardless of whether a participant took any investigational medicinal product (IMP).
Groups:
- ABS eMDPI: Participants received 90 mcg of ABS via eMDPI (sitting on the upper part of the device for the purposes of detecting and storing usage information), 1 to 2 inhalations every 4 hours, as needed for 12 weeks. ABS eMDPI was a rescue/reliever agent that included an eModule on top of the approved PROAIR RESPICLICK® inhaler. Participants were allowed to continue use of other asthma and non-asthma medications as advised by their physician without changes unless deemed necessary by their physician.
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 318
  Male | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99
  Not Hispanic or Latino | 298
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 74
  White | 313
  Other | 2
Number of Asthma Exacerbations in the Past 12 Months [Mean (Standard Deviation); unit: exacerbations] — Population: Here, 'number analyzed' signifies number of participants with asthma exacerbations.
  exacerbations
    number analyzed (Participants) | 394
    (all) | 1.5 (1.29)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Asthma Exacerbation (CAE) Rate: Percentage of Participants Who Experienced at Least 1 Moderate or Severe CAE
Description: CAE was an occurrence of either severe CAE or moderate CAE. Severe CAE was defined as a CAE that involved worsening asthma such that the treating physician elected to administer prednisone (or equivalent glucocorticoid treatment) at least 10 milligrams (mg) prednisone equivalent above Baseline, for at least 3 days; and an unscheduled provider visit such as an office visit, urgent care visit, emergency care visit, or hospitalization.
  Moderate CAE was defined as a CAE that involved worsening asthma such that the treating physician elected to administer prednisone (or equivalent glucocorticoid treatment) at least 10 mg prednisone equivalent above Baseline, for at least 3 days, or an unscheduled provider visit such as an office visit, urgent care visit, emergency care visit, or hospitalization associated with an increase in asthma therapy that did not qualify for severe CAE as defined above.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP.
Measure: Number; unit: percentage of participants
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 397
percentage of participants | 17

2. Primary Outcome: Total Number of Inhalations in the Days Preceding the Peak of a Severe CAE
Description: Severe CAE was defined as a CAE that involved worsening asthma such that the treating physician elected to administer prednisone (or equivalent glucocorticoid treatment) at least 10 mg prednisone equivalent above Baseline, for at least 3 days; and an unscheduled provider visit such as an office visit, urgent care visit, emergency care visit, or hospitalization. Total number of inhalations taken in 1 day (that is, the 24-hour period on the day prior to the date of the CAE symptom peak) and at 3, 5, 7, 10, 14, and 21 days preceding the date of the severe CAE symptom peak were reported.
Time Frame: Baseline to Week 12
Population: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP. Here, 'overall number of participants analyzed' signifies number of participants experiencing at least 1 severe CAE. Here, 'number analyzed' signifies participants who reported albuterol use in specified time interval.
Measure: Mean (Standard Deviation); unit: inhalations
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 37
inhalations
  Day 1 prior to CAE: number analyzed (Participants) | 31
  Day 1 prior to CAE | 5.9 (7.95)
  Day 3 prior to CAE: number analyzed (Participants) | 28
  Day 3 prior to CAE | 6.1 (9.93)
  Day 5 prior to CAE: number analyzed (Participants) | 26
  Day 5 prior to CAE | 3.6 (2.89)
  Day 7 prior to CAE: number analyzed (Participants) | 23
  Day 7 prior to CAE | 4.0 (2.61)
  Day 10 prior to CAE: number analyzed (Participants) | 26
  Day 10 prior to CAE | 4.5 (4.24)
  Day 14 prior to CAE: number analyzed (Participants) | 28
  Day 14 prior to CAE | 3.2 (1.87)
  Day 21 prior to CAE: number analyzed (Participants) | 22
  Day 21 prior to CAE | 4.0 (3.06)

3. Primary Outcome: Number of Days Prior to the Peak of a Severe CAE When Albuterol Use Increased
Description: Severe CAE was defined as a CAE that involved worsening asthma such that the treating physician elected to administer prednisone (or equivalent glucocorticoid treatment) at least 10 mg prednisone equivalent above Baseline, for at least 3 days; and an unscheduled provider visit such as an office visit, urgent care visit, emergency care visit, or hospitalization. Number of days prior to the peak of a severe CAE when albuterol use first increased to greater than (>) 4, >12, and >20 inhalations was reported. Participants were counted in more than 1 category (that is, all of the >20 inhalation participants were also counted in the >12 category, and in the >4 category).
Time Frame: Baseline to Week 12
Population: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP. Here, 'overall number of participants analyzed'= number of participants experiencing at least 1 severe CAE. 'Number analyzed'= participants who had any single day prior to CAE where their albuterol use exceeded 4, 12, or 20 inhalations in that day.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 37
days
  Albuterol use >4 inhalations: number analyzed (Participants) | 29
  Albuterol use >4 inhalations | 39.3 (26.79)
  Albuterol use >12 inhalations: number analyzed (Participants) | 9
  Albuterol use >12 inhalations | 40.3 (26.95)
  Albuterol use >20 inhalations: number analyzed (Participants) | 6
  Albuterol use >20 inhalations | 34.0 (30.84)

4. Primary Outcome: Number of Albuterol Uses in the 24 Hours Preceding a Severe CAE
Description: Severe CAE was defined as a CAE that involved worsening asthma such that the treating physician elected to administer prednisone (or equivalent glucocorticoid treatment) at least 10 mg prednisone equivalent above Baseline, for at least 3 days; and an unscheduled provider visit such as an office visit, urgent care visit, emergency care visit, or hospitalization. Number of albuterol inhalations used in the 24 hours preceeding a severe CAE is reported.
Time Frame: Baseline to Week 12
Population: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP. Here, 'overall number of participants analyzed' signifies number of participants who experienced at least 1 severe CAE and reported albuterol use in the 24 hours preceding a severe CAE.
Measure: Mean (Standard Deviation); unit: inhalations
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 31
inhalations | 5.9 (7.95)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by investigator. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to week 12
Population: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 397
Participants
  Any AEs | 127
  Severe AEs | 41
  Treatment-related AEs | 2
  Treatment-related severe AE | 0
  Serious AEs | 6
  AEs leading to discontinuation from study | 2
  CAE related AEs | 73
  Device-related AEs | 3
  AEs leading to death | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP.
Arm/Group | ABS eMDPI
All-Cause Mortality (participants affected / at risk) | 0/397
Serious Adverse Events (participants affected / at risk) | 6/397
Other Adverse Events (participants affected / at risk) | 68/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABS eMDPI (N=397)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABS eMDPI (N=397)
Asthma (Respiratory, thoracic and mediastinal disorders) | 68 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT02969408/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT02969408/SAP_001.pdf